CLINICAL TRIAL: NCT05996926
Title: Diagnostic Correlation Between Saline Infused Sonohystrography and Three Dimensional Transvaginal Ultrasound in the Assessment of Cesarean Section Scar Defect. A Study of a Diagnostic Test Accuracy
Brief Title: Diagnostic Accuracy of Saline Sonohystrography vs. 3D Transvaginal Ultrasound for Cesarean Scar Defect Assessment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Israa Bahaa Hassan Sherif, Resident of Obstetrics and Gynecology, Nile specialized Hospital, Egypt, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: FMASU MD25/2021
Record Dates: First submitted 2023-08-03; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Cesarean Scar Defects; Cesarean Section Complications; Uterine Scar Dehiscence; Vaginal Birth After Cesarean; Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-Dimensional Transvaginal Ultrasound (3D TVS) (Experimental): In this study, Three-Dimensional Transvaginal Ultrasound will be employed as one of the interventions to evaluate Cesarean Scar Defects (CSD) and associated complications in symptomatic patients with a history of cesarean section.
  A specialized ultrasound machine (Samsung WS80A) equipped with a transvaginal 2-11 MHz probe will be used for the Three-Dimensional Transvaginal Ultrasound examination. The examination will be conducted in the 1st half of the menstrual cycle. The ultrasound probe will be introduced into the posterior fornix of the vagina to capture three-dimensional images of the uterus and scar area. The examiner will identify and measure the characteristics of the Cesarean Scar Defects (CSD), including length, depth, width, volume, residual myometrial thickness, adjacent myometrial thickness, and presence of any branches.
  Interventions: Diagnostic Test: Three-Dimensional Transvaginal Ultrasound (3D TVS)
- Saline-Infused Sonography (Sonohystrography) (Experimental): The Sonohystrography will be performed using a Toshiba ECCO CEE SSA-340A ultrasound equipment with a 7.5 MHz transvaginal probe. A sterile vaginal speculum will be inserted, the cervix cleansed with an antiseptic solution, and a thin Foley's catheter inserted into the cervical os. Sterile saline solution will be infused into the uterus through the catheter to distend the uterine cavity. The examiner will use the ultrasound probe to visualize and assess the uterine cavity, focusing on identifying and measuring Cesarean Scar Defects (CSD) characteristics, including depth, width, volume, and myometrial thickness.
  Interventions: Diagnostic Test: Saline-Infused Sonography (Sonohystrography)

INTERVENTIONS:
Diagnostic Test: Three-Dimensional Transvaginal Ultrasound (3D TVS) — In this study, Three-Dimensional Transvaginal Ultrasound will be employed as one of the interventions to evaluate Cesarean Scar Defects (CSD) and associated complications in symptomatic patients with a history of cesarean section.
  Procedure: A specialized ultrasound machine (Samsung WS80A) equipped with a transvaginal 2-11 MHz probe will be used for the Three-Dimensional Transvaginal Ultrasound examination. The examination will be conducted in the 1st half of the menstrual cycle. The ultrasound probe will be introduced into the posterior fornix of the vagina to capture three-dimensional images of the uterus and scar area. The examiner will identify and measure the characteristics of the Cesarean Scar Defects (CSD), including length, depth, width, volume, residual myometrial thickness, adjacent myometrial thickness, and presence of any branches.
  Arms: Three-Dimensional Transvaginal Ultrasound (3D TVS)
Diagnostic Test: Saline-Infused Sonography (Sonohystrography) — The Sonohystrography will be performed using a Toshiba ECCO CEE SSA-340A ultrasound equipment with a 7.5 MHz transvaginal probe. A sterile vaginal speculum will be inserted, the cervix cleansed with an antiseptic solution, and a thin Foley's catheter inserted into the cervical os. Sterile saline solution will be infused into the uterus through the catheter to distend the uterine cavity. The examiner will use the ultrasound probe to visualize and assess the uterine cavity, focusing on identifying and measuring Cesarean Scar Defects (CSD) characteristics, including depth, width, volume, and myometrial thickness.
  Arms: Saline-Infused Sonography (Sonohystrography)

SUMMARY:
To compare accuracy of three dimensional transvaginal ultrasound versus the "gold standard" saline infused sonography for assessing the characteristics, frequency and appearance of caesarean scar defects in symptomatic patients with a history of cesarean section.

DETAILED DESCRIPTION:
Cesarean section (CS) is a frequently performed surgical procedure in obstetric practice. With a significant number of women undergoing this procedure annually, studying its impact on future reproductive capacity has become increasingly important.

The prevalence of cesarean deliveries is rising and constitutes about one-third of all births in both the USA and Italy. As the use of cesarean delivery increases, so do the associated complications, including cesarean scar pregnancy, morbidly adherent placenta, and Cesarean section scar dehiscence and rupture.

Cesarean scar defects (CSD) are described using various terms (pouch, niche, or isthmocoele) and are characterized by thinning of the myometrium or a uterine scar dehiscence, often appearing as a triangular shape within the endometrial cavity.

The exact prevalence of symptomatic Cesarean scar defects varies due to factors like population differences and lack of standardized criteria. Clinical presentations of Cesarean scar defects range from no symptoms to abnormal uterine bleeding, infertility, dyspareunia, and pelvic pain.

Women with a history of Cesarean section are considered high-risk during pregnancy and require specialized assessments to ensure scar integrity. Saline-infused sonography (Sonohystrography) is effective for demonstrating caesarean niches, although transvaginal ultrasound (TVS) is more accessible and commonly used.

Experts generally agree that a niche should be defined by an indentation at the CS scar site with a depth of at least 2 mm, and it can be classified as simple, simple with one branch, or complex with multiple branches. Additional measurements, such as the distances between the niche and the vesicovaginal fold, are useful for surgical planning.

Given the increasing frequency of cesarean deliveries, healthcare providers will encounter related complications more frequently. Cesarean scar defects are common yet often go undiagnosed. Encouraging vaginal birth after cesarean (VBAC) can help reduce cesarean rates and raise questions about future obstetric practices, especially in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 45 years
* Previous 1-3 cesarean sections
* The duration from the last cesarean section ranging from 6 months to 5 years.

Exclusion Criteria:

* Pregnancy (Positive pregnancy test)
* Recent pelvic infection.
* Active pelvic infection.
* Recent surgery on the tubes or the uterus.
* Active vaginal bleeding.
* Menstruation.
* Suspected malignancy.
* Intrauterine device in situ.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women aged between 20 and 45 years with a history of 1 to 3 previous cesarean sections (CS) and a duration of time since the last CS ranging from 6 months to 5 years will be eligible for enrollment in this study.
Enrollment: 72 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Cesarean Scar Defect Assessment Using 3D TVS | Intraoperatively
  This outcome measure aims to evaluate the diagnostic accuracy of three-dimensional transvaginal ultrasound (3D TVS) as measurement tools in assessing Cesarean Scar Defects (CSD) and associated complications among symptomatic patients with a history of cesarean section. The assessment will involve identifying, classifying, and measuring Cesarean Scar Defects (CSD) characteristics using these specific measurement techniques.
Diagnostic Accuracy of Cesarean Scar Defect Assessment Using Saline-Infused Sonography | Intraoperatively
  This outcome measure aims to evaluate the diagnostic accuracy of saline-infused sonography (Sonohystrography) as measurement tools in assessing Cesarean Scar Defects (CSD) and associated complications among symptomatic patients with a history of cesarean section. The assessment will involve identifying, classifying, and measuring Cesarean Scar Defects (CSD) characteristics using these specific measurement techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be available upon a reasonable request.
Supporting Information: Study Protocol
Time Frame: One you after the end of the study